CLINICAL TRIAL: NCT03805178
Title: Lung Transplant Plasmapheresis (PLEX)/Belatacept/Carfilzomib Protocol for Treatment of Antibody Mediated Rejection (AMR) and Desensitization
Brief Title: Lung Transplant Plasmapheresis/Belatacept/Carfilzomib for Antibody Mediated Rejection and Desensitization
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not activated at Duke
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00101289; IM103-407 (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Lung Transplant Rejection; Antibody-mediated Rejection
MeSH Terms: interventions — Abatacept; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rejection post-transplant (Experimental): Treatment with Belatacept and Carfilzomib for subjects who show evidence of antibody-mediated rejection (AMR) following lung transplantation.
  Interventions: Drug: Belatacept; Drug: Carfilzomib
- Pre-transplant desensitization (Experimental): Treatment with Belatacept and Carfilzomib for subjects with elevated human leukocyte antigen (HLA) antibodies prior to lung transplantation.
  Interventions: Drug: Belatacept; Drug: Carfilzomib

INTERVENTIONS:
Drug: Belatacept — Initial phase: 10 mg/kg on days 0 and 4, and again at weeks 2 and 4. Maintenance phase: 10 mg/kg every month beginning 4 weeks after completion of the initial phase.
  No dosage adjustments required for renal or hepatic impairment. No known drug interactions for usual post-transplant medication regimen.
  Other Names: Nulojix
Drug: Carfilzomib — 20mg/m2 Plasmapheresis
  Other Names: Kyprolis

SUMMARY:
Antibody mediated rejection (AMR) post transplant contributes to poor long term outcomes after lung transplantation. Additionally, high antibodies detected pre transplant in candidates limit donor availability for lung transplant. This proposal would include belatacept in a multi-therapy regimen. Open label study with two patient cohorts for safety and efficacy of belatacept in a multi-modal protocol. The two patient cohorts are an AMR post-transplant cohort and pre-transplant desensitization cohort. A total of 10 patients will be enrolled.The primary objection is drug tolerability and secondary objectives are antibody measurements and allograft function.

DETAILED DESCRIPTION:
Antibody mediated rejection (AMR) post transplant contributes to poor long term outcomes after lung transplantation. Additionally, high antibodies detected pre transplant in candidates limit donor availability for lung transplant. Multimodal therapies with rituximab, intravenous immunoglobulin, plasmapheresis and proteasome inhibitors have not significantly altered the antibodies in these patients. Belatacept targets the T and B cell interaction such that it represents a novel therapeutic strategy. This proposal would include belatacept in a multi-therapy regimen.

This is an open label study with two patient cohorts for safety and efficacy of belatacept in a multi-modal protocol. The two patient cohorts are an AMR post-transplant cohort and pre-transplant desensitization cohort. A total of 10 patients will be enrolled.The primary objection is drug tolerability and secondary objectives are antibody measurements and allograft function.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the AMR post-transplant cohort

* Positive DSAs and allograft dysfunction defined by changes in pulmonary physiology, gas exchange, radiological features or deteriorating functional performance that is highly suspicious for AMR
* Recipient is Epstein-Barr virus positive (EBV+) by serology
* Ability to provide signed and dated IRB approved written consent in accordance with regulatory and institutional guidelines prior to any protocol-related procedure

Inclusion criteria for the pre-transplant desensitization cohort

* Elevated HLA antibodies (defined as MFI >1000) such that the calculated panel reactive antibodies are >60%
* At least 2 HLA antibodies with Mean Fluorescent Intensity (MFI) <10,000 and at least 2 HLA antibodies with MFI <5,000 on undiluted serum that do not demonstrate an increase in MFI with dilution at 1:16 (no evidence of a prozone effect).
* EBV+ by serology
* Clinically stable defined by not on invasive mechanical ventilation, extracorporeal membrane oxygenation support or other invasive life support requiring ICU level of care
* Ability to provide signed and dated IRB approved written consent in accordance with regulatory and institutional guidelines prior to any protocol-related procedure

Exclusion criteria for both AMR post-transplant cohort and pre-transplant cohort

* Active systemic infection
* Allergy to carfilzomib or belatacept
* Known malignancy in the previous 2 years except for non-melanomatous skin cancer
* Pregnancy
* Inability to commit to complete treatment protocol at Duke as all procedures must be completed at Duke
* Prisoners or those who are compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of drug side effects | Within 28 days of last administration of study drugs
  Drug tolerability with respect to freedom from drug side effects measured using descriptive statistics
Occurrence of infection | Within 28 days of last administration of study drugs
  Drug tolerability with respect to freedom from infection measured using descriptive statistics
Occurrence of malignancy | Within 28 days of last administration of study drugs
  Drug tolerability with respect to freedom from malignancy measured using descriptive statistics

SECONDARY OUTCOMES:
Number of subjects in the AMR cohort with resolution of at least one donor specific human leukocyte antigen (HLA) antibody (DSA) | Within 4 weeks of completion of treatment
  Descriptive statistical report of number of subjects who had resolution of at least one DSA measured by absolute Mean Fluorescent Intensity (MFI) change and log change using pre and post treatment values for each antibody.
Number of subjects in the AMR cohort with improvement or stabilization of lung function as measured by spirometry data | Within 4 weeks of completion of treatment
  Pulmonary function (spirometry) data will track forced vital capacity (FVC), forced expiratory volume (FEV1) and forced expiratory flow (FEF) 25-75%. Changes in spirometry will be reported as stabilized, improved or worsened based on comparison of baseline spirometry values obtained prior to treatment plan with serial spirometric testing performed at specified intervals in treatment plan.
Number of subjects in the AMR cohort with improvement in oxygenation as measured by Liters/min oxygen at rest | Within 4 weeks of completion of treatment
  Gas exchange will be reported as no change, worsening exchange or improving exchange based on comparison of resting oxygen requirements before and following treatment plan.
Number of subjects in the AMR cohort with decrease in DSA by one log | Within 4 weeks of completion of treatment
  Descriptive statistical report of number of subjects who had a decrease in DSA measured by absolute Mean Fluorescent Intensity (MFI) change and log change using pre and post treatment values for each antibody.
Number of subjects in the AMR cohort with elimination of DSA at 1:16 dilution | Within 4 weeks of completion of treatment
  Descriptive statistical report of number of subjects who had elimination of DSA at 1:16 dilution measured by absolute Mean Fluorescent Intensity (MFI) change and log change using pre and post treatment values for each antibody.
Number of subjects in the transplant desensitization cohort with decrease in non-DSA HLA antibodies by one log | Within 4 weeks of completion of treatment
  Descriptive statistical report of number of subjects who had a decrease in non-DSA HLA antibodies measured by absolute Mean Fluorescent Intensity (MFI) change and log change using pre and post treatment values for each antibody.
Number of subjects in the transplant desensitization cohort with elimination of non-DSA HLA antibodies at 1:16 dilution | Within 4 weeks of completion of treatment
  Descriptive statistical report of number of subjects who had elimination of non-DSA HLA antibodies at 1:16 dilution measured by absolute Mean Fluorescent Intensity (MFI) change and log change using pre and post treatment values for each antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Snyder, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No